CLINICAL TRIAL: NCT01128946
Title: Comparison of Enamel Remineralization Potential of Dentifrices Incorporating Different Fluoride Salts Using an in Situ Caries Model
Brief Title: Enamel Remineralization Potential of Dentifrices in Situ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: T3500690
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2013-11-04 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Dental Caries
Keywords: Enamel remineralization; Fluoride; caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fluoride Toothpaste 1 (Experimental): Fluoride toothpaste containing sodium fluoride (NaF)
  Interventions: Drug: NaF
- Fluoride Toothpaste 2 (Experimental): Fluoride toothpaste containing stannous fluoride (SnF) and NaF.
  Interventions: Drug: NaF; Drug: SnF
- Fluoride Toothpaste 3 (Experimental): Fluoride toothpaste containing sodium monofluorophosphate (NaMFP) and NaF.
  Interventions: Drug: NaF; Drug: NaMFP
- Reference Dentifrice (Active Comparator): Low fluoride toothpaste containing NaF
  Interventions: Drug: NaF

INTERVENTIONS:
Drug: NaF — Fluoride toothpaste containing sodium fluoride as 1450 parts per million (ppm) F, 675 ppmF, 450 ppmF, 350ppmF.
Drug: SnF — Fluoride toothpaste containing stannous fluoride (1100 ppmF)
  Arms: Fluoride Toothpaste 2
Drug: NaMFP — Fluoride toothpaste containing sodium monofluorophosphate (1000 ppmF)
  Arms: Fluoride Toothpaste 3

SUMMARY:
This study will use an oral in-situ caries model to study remineralization of enamel due to the action of different combinations of fluoride salts delivered from dentifrices.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical or oral health.
* No current active caries or periodontal disease that may compromise the study or health of the subject.
* All restorations in a good state of repair
* Currently wearing a removable mandibular partial denture with sufficient room in the posterior buccal flange area to accomodate two enamel specimens required dimensions 12 x 7 mm.
* Willing to have their denture modified to accomodate enamel test specimens
* Willing and capable of wearing removable mandibular partial dentures 24 hours per day during the treatment periods.
* Salivary flow rate in the range of normal values (unstimulated whole saliva flow rate greater than or equal to 0.2 mL/ minute; gum base stimulated whole saliva flow rate greater than or equal to 0.8 mL/minute.

Exclusion Criteria:

* Individuals currently taking antibiotics, or who have taken antibiotics within 30 days prior to the first treatment visit.
* Current active caries or periodontal disease that may compromise the study or health of the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Two to three days before the start of each treatment period, participants received a professional dental cleaning of their natural teeth, then brushed with the study wash out toothpaste and toothbrush.
Groups:
- Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F: Participants brushed their natural teeth twice daily, for one timed minute, with 1.5 gram (g) NaF toothpaste (1450ppmF as NaF), followed by rinsing with 15 milliliters (mL) water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days with instructions to not brush the enamel specimens. Participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF: Participants brushed their natural teeth twice daily, for one timed minute with 1.5g NaMFP and NaF toothpaste (1000ppmF as NaMFP and 450ppmF as NaF), followed by rinsing with 15 mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days with instructions to not brush the enamel specimens. Participants wore their partial dentures 24-hours a day, except when cleaning their dentures
- Strontium Fluoride (SnF)/NaF Toothpaste (1450ppmF: Participants brushed their natural teeth twice daily, for one timed minute, with 1.5 g SnF toothpaste (1100ppmF as SnF and 350ppmF as NaF), followed by rinsing with 15mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days with instructions to not brush the enamel specimens. Participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- NaF Toothpaste (675ppmF: Participants brushed their natural teeth twice daily, for one timed minute with NaF toothpaste (675ppmF as NaF), followed by rinsing with 15mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days with instructions to not brush the enamel specimens. Participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
Period: Period I
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF | Strontium Fluoride (SnF)/NaF Toothpaste (1450ppmF | NaF Toothpaste (675ppmF
Started | 20 | 21 | 21 | 21
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Period: Period II
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF | Strontium Fluoride (SnF)/NaF Toothpaste (1450ppmF | NaF Toothpaste (675ppmF
Started | 20 (Due to crossover design, different set of participants received this treatment compared to Period I) | 20 (Due to crossover design, different set of participants received this treatment compared to Period I) | 20 (Due to crossover design, different set of participants received this treatment compared to Period I) | 20 (Due to crossover design, different set of participants received this treatment compared to Period I)
Completed | 20 | 19 | 20 | 19
Not Completed | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Period III
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF | Strontium Fluoride (SnF)/NaF Toothpaste (1450ppmF | NaF Toothpaste (675ppmF
Started | 20 (Due to crossover design, different set of participants received this treatment compared to Period II) | 19 (Due to crossover design, different set of participants received this treatment compared to Period II) | 20 (Due to crossover design, different set of participants received this treatment compared to Period II) | 19 (Due to crossover design, different set of participants received this treatment compared to Period II)
Completed | 19 | 19 | 20 | 19
Not Completed | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Period: Period IV
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF | Strontium Fluoride (SnF)/NaF Toothpaste (1450ppmF | NaF Toothpaste (675ppmF
Started | 19 (Due to crossover design,different set of participants received this treatment compared to Period III) | 20 (Due to crossover design,different set of participants received this treatment compared to Period III) | 19 (Due to crossover design,different set of participants received this treatment compared to Period III) | 19 (Due to crossover design,different set of participants received this treatment compared to Period III)
Completed | 19 | 20 | 19 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All randomized participants
Arm/Group | Overall
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 35
Region of Enrollment [Number; unit: Participants]
  United States | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Microhardness Recovery (%SMHR) of Enamel Specimens Exposed to NaF Toothpaste (1450ppmF) and SnF/NaF Toothpaste (1450ppmF)
Description: SMH test was used to assess mineral status of partially demineralized enamel specimens using Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening/demineralization, while decrease in the indentation represents rehardening/ remineralization of enamel surface. Percent SMH recovery was calculated from indentation values of enamel specimens at baseline(B), after intra-oral exposure(R) and after in-vitro demineralization(D) using formula: [(D-R)/(D-B)]*100.
Time Frame: Baseline to 14 days
Population: Per Protocol (PP) population: All randomized participants, who received at least one dose of study treatment and with at least one post-baseline efficacy assessment but did not have any major protocol violations. Missing data was not imputed. Due to drop outs, there were differences in number of participants (N) per treatment group.
Measure: Mean (Standard Error); unit: Percentage of SMHR
Groups:
- NaF Toothpaste (1450ppmF): Participants brushed their natural teeth twice daily, for one timed minute, with 1.5 g NaF toothpaste (1450ppmF as NaF), followed by rinsing with 15 mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days with instructions to not brush the enamel specimens. Participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- SnF/NaF Toothpaste (1450ppmF): Participants brushed their natural teeth twice daily, for one timed minute, with 1.5 g SnF toothpaste (1100ppmF as SnF and 350ppmF as NaF), followed by rinsing with 15mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days with instructions to not brush the enamel specimens. Participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
Arm/Group | NaF Toothpaste (1450ppmF) | SnF/NaF Toothpaste (1450ppmF)
Number analyzed (Participants) | 78 | 79
Percentage of SMHR | 40.94 (1.930) | 17.88 (1.924)
Statistical Analysis 1: Comparison: NaF Toothpaste (1450ppmF) vs SnF/NaF Toothpaste (1450ppmF); Null hypothesis considered population means for treatments in comparison, to be equal with respect to percent SMH recovery. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 23.06, 95% CI 2-sided [19.63 to 26.48] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment

2. Secondary Outcome: %SMHR of Enamel Specimens Exposed to NaF Toothpaste (1450ppmF), SnF/NaF Toothpaste (1450ppmF), NaMFP/NaF Toothpaste (1450ppmF) and NaF Toothpaste (675ppmF)
Description: SMH test was used to assess mineral status of partially demineralized enamel specimens using Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening/demineralization, while decrease in the indentation represents rehardening/ remineralization of enamel surface. Percent SMH recovery was calculated from indentation values of enamel specimens at baseline(B), after intra-oral exposure(R) and after in-vitro demineralization(D) using formula: [(D-R)/ (D-B)]*100.
Time Frame: Baseline to 14 days
Population: PP population: All randomized participants, who received at least one dose of study treatment and with at least one post-baseline efficacy assessment but did not have any major protocol violations. Missing data was not imputed. Due to drop outs, there were differences in number of participants (N) per treatment group
Measure: Mean (Standard Error); unit: Percentage
Groups:
- NaMFP/NaF Toothpaste (1450ppmF): Participants brushed their natural teeth twice daily, for one timed minute with 1.5g NaMFP and NaF toothpaste (1000ppmF as NaMFP and 450ppmF as NaF), followed by rinsing with 15 mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days with instructions to not brush the enamel specimens. Participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- NaF Toothpaste (675ppmF): Participants brushed their natural teeth twice daily, for one timed minute with NaF toothpaste (675ppmF as NaF), followed by rinsing with 15mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days with instructions to not brush the enamel specimens. Participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
Arm/Group | NaF Toothpaste (1450ppmF) | NaMFP/NaF Toothpaste (1450ppmF) | SnF/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF)
Number analyzed (Participants) | 78 | 78 | 79 | 76
Percentage | 40.94 (1.93) | 30.19 (1.932) | 17.88 (1.924) | 28.74 (1.943)
Statistical Analysis 1: Comparison: NaF Toothpaste (1450ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 10.75, 95% CI 2-sided [7.33 to 14.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 12.20, 95% CI 2-sided [8.74 to 15.67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs SnF/NaF Toothpaste (1450ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 12.31, 95% CI 2-sided [8.90 to 15.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4070, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 1.46, 95% CI 2-sided [-2.00 to 4.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: SnF/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = -10.85, 95% CI 2-sided [-14.30 to -7.40] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Enamel Fluoride Uptake Upon Exposure to NaF Toothpaste (1450ppmF), SnF/NaF Toothpaste (1450ppmF), NaMFP/NaF Toothpaste (1450ppmF) and NaF Toothpaste (675ppmF)
Description: Enamel fluoride uptake was determined using the microdrill enamel biopsy technique. The amount of fluoride uptake by enamel was calculated based on the amount of fluoride (F) divided by the area of the enamel cores. The difference between treatments was calculated with respect to fluoride uptake by enamel.
Time Frame: Baseline to 14 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: micrograms (μg)*F/centimeters(cm)^2]
Arm/Group | NaF Toothpaste (1450ppmF) | NaMFP/NaF Toothpaste (1450ppmF) | SnF/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF)
Number analyzed (Participants) | 78 | 78 | 79 | 76
micrograms (μg)*F/centimeters(cm)^2] | 22.23 (0.853) | 13.54 (0.854) | 9.13 (0.850) | 14.31 (0.861)
Statistical Analysis 1: Comparison: NaF Toothpaste (1450ppmF) vs SnF/NaF Toothpaste (1450ppmF); Null hypothesis considered population means for treatments in comparison, to be equal with respect to enamel fluoride uptake. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 13.21, 95% CI 2-sided [11.46 to 14.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste (1450ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 8.79, 95% CI 2-sided [7.04 to 10.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 8.03, 95% CI 2-sided [6.25 to 9.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs SnF/NaF Toothpaste (1450ppmF); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = 4.41, 95% CI 2-sided [2.66 to 6.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3942, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = -0.77, 95% CI 2-sided [-2.54 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: SnF/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period and subject (random effect); Adjusted Mean Difference = -5.18, 95% CI 2-sided [-6.95 to -3.41] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Arm/Group | NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | NaMFP/NaF Toothpaste (1450ppmF) | SnF/NaF Toothpaste (1450ppmF)
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 1/80 | 0/80
Other Adverse Events (participants affected / at risk) | 10/79 | 12/79 | 18/80 | 15/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF Toothpaste (1450ppmF) (N=79) | NaF Toothpaste (675ppmF) (N=79) | NaMFP/NaF Toothpaste (1450ppmF) (N=80) | SnF/NaF Toothpaste (1450ppmF) (N=80)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF Toothpaste (1450ppmF) (N=79) | NaF Toothpaste (675ppmF) (N=79) | NaMFP/NaF Toothpaste (1450ppmF) (N=80) | SnF/NaF Toothpaste (1450ppmF) (N=80)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 3 (4)
Gastrointestinal Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis Infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival Erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gingival Ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chapped Lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth Injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (4) | 1 (2) | 3 (3)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tongue Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning Sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve Compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.